CLINICAL TRIAL: NCT02800967
Title: Investigation of Beneficial Effects of Aronia Juice (Aronia Melanocarpa) and Dietary Polyphenols on the Activity of Thrombocytes as Well as Other Risk Factors Causing Cardio-vascular Diseases
Brief Title: The Effects of Aronia Juice Polyphenols on Cardiovascular Disease Risk
Acronym: AMARCord
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Belgrade (Other)
Collaborators: Clinical Hospital Center Zemun (Other)
Responsible Party: Principal Investigator, Maria Glibetic, Professor, PhD, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Bacchus_AMARCord_2013
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension; Overweight
Keywords: platelet activation; platelet aggregation; Aronia; flow cytometry; polyphenols; cardiovascular disease risk
MeSH Terms: conditions — Hypertension; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pure Aronia juice (Active Comparator): Participants will consume 100 ml of pure Aronia juice per day for 28 days
  Interventions: Dietary Supplement: Pure Aronia juice
- Aronia juice-based beverage (Active Comparator): Participants will consume 100 ml of Aronia juice-based beverage per day for 28 days.
  Interventions: Dietary Supplement: Aronia juice-based beverage
- Placebo beverage (Placebo Comparator): Participants will consume 100 ml of Placebo beverage per day for 28 days
  Interventions: Dietary Supplement: Placebo beverage

INTERVENTIONS:
Dietary Supplement: Pure Aronia juice — Pure Aronia juice with appx. polyphenols content of 1000 mg gallic acid equivalents/100ml
  Arms: Pure Aronia juice
Dietary Supplement: Aronia juice-based beverage — Aronia juice-based beverage with appx. polyphenols content of 250 mg gallic acid equivalents/100ml, obtained as a blend of ¼ vol. of pure Aronia juice and ¾ vol. of placebo beverage.
  Arms: Aronia juice-based beverage
Dietary Supplement: Placebo beverage — A polyphenol-free formulation with matched nutrient composition (sugars, vitamins, minerals) and similar sensory characteristics to active interventions
  Arms: Placebo beverage

SUMMARY:
The existing scientific evidence from both in vitro and clinical trials supports the notion that polyphenols can modulate platelet function. Beyond being central players in haemostasis and thrombosis, platelets have crucial roles in the development of atherosclerosis, mediated through their interactions with monocytes and endothelial cells. Disturbed platelet function correlates with other risk factors, including hypertension and obesity, and the progression of cardiovascular diseases (CVD), postulating platelets as rational targets in CVD prevention. Thus, the effects of polyphenols on disturbed platelet function would contribute to their pleiotropic beneficial effects of on cardiovascular health. Aronia juice is a rich source of polyphenols including anthocyanins, procyanidins, phenolic acids and flavonols. However, there is no clinical evidence on the effects of aronia juice consumption on platelet function and related CVD factors. The purpose of this study is to investigate the effects of Aronia juice polyphenols on platelet function and other CVD risk factors in subjects with moderate CVD risk.

DETAILED DESCRIPTION:
To investigate the effect of Aronia (Aronia melanocarpa L.) juice polyphenols on platelet function and other CVD risk factors a three-arm, crossover design, randomized, double-blind placebo-controlled clinical trial will be performed in apparently healthy subjects at moderate CVD risk.

Recruited participants will be randomly assigned to one of three interventions (pure Aronia juice, Aronia beverage or placebo beverage) in the first phase and followed by cross-over in second and third phase. Two-week run-in period with low intake of polyphenols will precede the start of the intervention, ie. the first intervention phase. During each of three intervention periods (phases) subjects will consume 100 ml of each intervention product daily for 28 days, with 28 days of wash out period between different phases.

Blood and urine samples will be taken at baseline, before and after 28 days after each intervention period. Platelet analyses by flow cytometry, biochemical analyses of plasma samples, full blood count, blood pressure and anthropometric measurements will be performed at each study visit.

During the first study visit, regardless the allocation, blood samples will be taken before and 2h after the consumption of first 100 ml of intervention product (performed at the experimental site) and the analysis of markers of platelet function, biochemical parameters (glucose, triglycerides, and uric acid) and blood pressure will be assessed.

Subjects will be instructed to avoid rich-sources of anthocyanins and procyanidins during the whole study. Dietary habits will be assessed by food frequency questionnaire (FFQ) performed 2 times at the beginning and at the end of the study and 24h-recall performed at the beginning and after each wash out period.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25-30 or
* Central obesity ie. WC≥80 cm (women) and ≥94 cm (man) or
* Normal (systolic blood pressure (SBP): 120-129; diastolic blood pressure(DBP): 80-84) or high normal (SBP:130-139; DBP:85-89) blood pressure

Exclusion Criteria:

* Smokers
* Diagnosed with CVD, history of stroke or CVD
* Diagnosis of type 2 diabetes mellitus on insulin therapy
* Very low or high blood pressure (<90/50)
* Pregnant or have been pregnant in the last 12 months or on oral contraceptives
* Gastrointestinal diseases
* Diagnosed with a long-term illness requiring active treatment, e.g. cancer, thyroid, adrenal, pituitary diseases
* On regularly prescribed medication known to have a profound effect on CVD risk factors (including statins)
* Non-steroidal anti-inflammatory drugs including creams
* Sufferers of asthma and/or hay-fever
* Known allergy to any of investigated polyphenol-rich food
* Regularly using antacids and laxatives (at least once a week)
* Unwillingness to discontinue specific dietary (other than vitamins and minerals) or herbal supplements less than one month prior to the start of the study and for the duration of the study
* Unwillingness to restrict oily fish consumption to 2 portions or less per week less than one month prior to the start of the study and for the duration of the study
* Taking paracetamol for more than one day during the intervention period and unwillingness to continue with the study intervention for an additional 48 hours if paracetamol is taken
* Blood donation within 16 weeks of the first study sample and who intend to donate blood less than 16 weeks after the last study sample
* Those who receive or plan to receive any type of immunization during the study period and those who have received an immunization within 4 weeks of the start of the study
* Parallel participation in another research project which involves dietary intervention (e.g. taking vitamin supplements) or sampling of blood that may increase the total volume taken above 470 mL in a 4 month period

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the percentage of P-selectin and glycoprotein IIbIIIa (GPIIbIIIa) positive platelets, percentage of platelet-monocyte and platelet-neutrophil aggregates, between baseline and endpoint within the intervention group vs. control group. | Baseline, 2 hours and 4 weeks
  Percentage of P-selectin and GPIIbIIIa positive platelets evaluated in total number of 20000 platelets, percentage of platelet-monocyte aggregates in 1000 monocytes and percentage of platelet-neutrophil aggregates in total 20000 neutrophils, all by flow cytometry, in non-treated blood samples and after ex vivo treatment of the whole blood with adenosine-diphosphate (0.5 μM and 20 μM)

SECONDARY OUTCOMES:
Changes in serum glucose levels between baseline and endpoint within the intervention group vs. control group. | Baseline, 2 hours and 4 weeks
  In 12h-fasting and 2h postprandial serum samples analysed by biochemical analyser.
Changes in serum cholesterol levels between baseline and endpoint within the intervention group vs. control group. | Baseline and 4 weeks
  Total cholesterol, LDL-cholesterol and HDL-cholesterol levels in 12h-fasting serum samples analysed by biochemical analyser
Changes in serum triglycerides levels between baseline and endpoint within the intervention group vs. control group. | Baseline, 2 hours and 4 weeks
  In 12h-fasting and 2h postprandial serum samples analysed by biochemical analyser
Changes in systolic and diastolic blood pressures between baseline and endpoint within the intervention group vs. control group. | Baseline, 2 hours and 4 weeks
  Mean of 3 x 2 consecutive office measurements performed within 30 min at each time point with professional OMRON device
Changes in body weight between baseline and 4 weeks within the intervention group vs. control group. | Baseline and 4 weeks
  Body weight will be measured by bio-impedance scale
Changes in waist circumference between baseline and 4 weeks within the intervention group vs. control group. | Baseline and 4 weeks
  Waist circumference will be measured by professional tape, according to the guidelines
Changes in body mass index between baseline and 4 weeks within the intervention group vs. control group. | Baseline and 4 weeks
  Body mass index will be calculated based on values obtained as body weight in kilograms divided by height in meters squared.
Changes in the percentage of body fat between baseline and 4 weeks within the intervention group vs. control group | Baseline and 4 weeks
  Body fat as percentage of total weight measured by bio-impedance instrument
Changes in the percentage of body water between baseline and 4 weeks within the intervention group vs. control group | Baseline and 4 weeks
  Body water as percentage of total weight measured by bio-impedance instrument
Changes in total body muscle mass between baseline and 4 weeks within the intervention group vs. control group | Baseline and 4 weeks
  Percentages of total body muscle mass in kilograms will be measured by bio-impedance instrument

OTHER OUTCOMES:
Changes in parameters of liver function between baseline and endpoint | Baseline and 4 weeks
  Aspartate transferase, alanine transferase , direct bilirubin, total bilirubin, gamma-glutamyl transferase , lactate dehydrogenase levels in 12h-fasting serum samples analysed by biochemical analyser
Changes in parameters of renal function between baseline and endpoint | Baseline and 4 weeks
  Urea and creatinine levels in 12h-fasting serum samples analysed by biochemical analyser
Changes in uric acid, iron and oxLDL level between baseline and endpoint within the intervention group vs. control group. | Baseline and 4 weeks
  In 12h-fasting serum samples analysed by biochemical analyser
Changes in full blood count between baseline and endpoint | Baseline and 4 weeks
Changes in total caloric intake and intake of total polyphenols | Baseline and 4 weeks
  Both caloric intake and intake of polyphenols will be assessed by standardized food-frequency questionnaire and 24-recall at baseline and after each wash-out period, based on data from Serbian Food Composition database. The agreements between two methods will also be assessed.
Changes in urine levels of major polyphenol metabolites between baseline and endpoint | Baseline, 2h and 4 weeks
  Measured in spot urine of total morning void by liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Maria Glibetic, Principal Investigator — University of Belgrade
Locations (1):
- Centre of Research Excellence in Nutrition and Metabolism, Institute for Medical Research, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stojkovic L, Zec M, Zivkovic M, Bundalo M, Boskovic M, Glibetic M, Stankovic A. Polyphenol-Rich Aronia melanocarpa Juice Consumption Affects LINE-1 DNA Methylation in Peripheral Blood Leukocytes in Dyslipidemic Women. Front Nutr. 2021 Jun 17;8:689055. doi: 10.3389/fnut.2021.689055. eCollection 2021. PMID 34222308